CLINICAL TRIAL: NCT00161993
Title: Prospective Open-Label Study of Pharmacokinetics, Efficacy and Safety of Immune Globulin Intravenous (Human), 10% TVR Solution in Patients With Hypo- or Agammaglobulinemia
Brief Title: Safety, Pharmacokinetic and Efficacy Study of a 10% Triple Virally Reduced Intravenous Immune Globulin Solution in Patients With Primary Immunodeficiency (Hypo- or Agammaglobulinemia)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 160001
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Primary Immunodeficiency Diseases (PID); Agammaglobulinemia; Hypogammaglobulinemia
Keywords: Gammaglobulin
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Agammaglobulinemia | interventions — gamma-Globulins; Solutions; Solvents; Detergents

INTERVENTIONS:
Drug: Immune Globulin Intravenous (Human), 10% TVR (Triple Virally Reduced) Solution
Drug: Gammagard S/D (Solvent/Detergent)

SUMMARY:
The purpose of this study is to determine the pharmacokinetics, efficacy and safety of Immune Globulin Intravenous (Human), 10% TVR (Triple Virally Reduced) Solution in subjects with primary immunodeficiency (PID) manifesting as hypo- or agammaglobulinemia. Subjects are treated every 21 days and receive a total of 12 infusions: for the first 3 infusions subjects receive GAMMAGARD S/D to ensure a steady-state and to acquire data with a licensed product; for the remaining 9 infusions subjects receive IGIV, 10% TVR Solution.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible for study entry if they:

* are at least 18 years old
* have a form of primary immunodeficiency (PID) as described by Rosen et al, 1999 16 manifesting as agammaglobulinemia (X-linked) or hypogamma-globulinemia (common variable immunodeficiency), requiring immunoglobulin replacement therapy
* have had regular treatment for at least three months with either intravenous immunoglobulin preparations or immunoglobulin preparations for intramuscular use given subcutaneously
* have serum IgG levels greater than or equal to 5 g/L as determined by the local laboratory at screening
* if female of childbearing potential, agree to employ adequate birth control measures during the study
* have given written informed consent

Exclusion Criteria:

Subjects will not be eligible for study entry if they:

* had severe adverse reactions to treatment with immunoglobulin preparations during the last three treatments before inclusion into the study
* suffer from documented selective IgA deficiency with antibodies against IgA
* have an acute infection that requires intravenous antibiotic treatment (Last treatment day should be seven days before study entry.)
* are known to be infected with HIV, HCV, or HBV
* are at high risk of contracting blood-borne viral infections through parenteral drug abuse or life style
* suffer from congestive heart failure and receive on-demand treatment with furosemide
* show renal dysfunction defined as serum creatinine greater than or equal to 1.5 mg/dL at baseline visit
* received another investigational drug in the three weeks preceding study entry
* in case of females, are pregnant or nursing mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2002-06-13 (Actual); Primary Completion 2003-09-24 (Actual); Study Completion 2003-09-24 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Trough levels of total immunoglobulin G (IgG) after treatment with Immune Globulin Intravenous (Human), 10% Triple Virally Reduced Solution (IGIV, 10% TVR Solution) | 21 days after each infusion (i.e., before the next infusion) of the study drug and at the last visit

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (6):
- Finland (2):
  - Tampere University Hospital, Tampere
  - Turku University Central Hospital, Turku
- Sweden (4):
  - SU/Sahlgrenska, Gothenburg
  - University Hospital Lund, Lund
  - University Hospital MAS, Malmo
  - Sundsvall Hospital, Sundsvall